CLINICAL TRIAL: NCT00006162
Title: Interventions to Reduce Diabetic Risk in Japanese Americans
Brief Title: Lifestyle Interventions to Reduce Diabetes Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: fujimotow (completed); 1R01DK048152 (NIH)
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Glucose Intolerance; Diabetes Mellitus, Type 2
Keywords: low fat diet; aerobic exercise; impaired glucose tolerance; Japanese Americans; metabolic risk factors
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Exercise; Diet

INTERVENTIONS:
Behavioral: exercise and diet

SUMMARY:
Type 2 diabetes is more frequent in Japanese Americans than in Japan or the U.S. non-Hispanic white population. This appears to be due to the effects of ''westernization'' to bring out metabolic changes that lead to diabetes. This study will look at whether increased physical activity and dietary changes will reduce or prevent the metabolic changes that lead to type 2 diabetes in Japanese Americans who have impaired glucose tolerance, a condition intermediate between normal glucose tolerance and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Japanese American
* Confirmed impaired glucose tolerance
* Able to fill out questionnaires

Exclusion Criteria:

* Significant exercise-restricting disease
* Poorly controlled hypertension
* Psychiatric disease or dementia
* Already on unusually restrictive diet
* Use of hypolipidemic drugs
* Use of tobacco
* Abnormal blood screening tests
* ECG evidence of ischemic heart disease at rest
* Abnormal maximal Bruce treadmill test

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-10; Study Completion 1999-04

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States